CLINICAL TRIAL: NCT00786266
Title: Sleep Enhancement Training Study for Novice Shiftworkers
Acronym: SETS-novice
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Christopher Alsten, PhD, Executive Vice President, Inner Health, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SETS-novice; R43NR010688 (NIH)
Record Dates: First submitted 2008-11-04; First posted 2008-11-06 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2010-06

CONDITIONS: Shift-Work Sleep Disorder
Keywords: shift-work; sleep; nurse; relaxation
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NIOSH shiftwork booklet (Active Comparator)
  Interventions: Behavioral: NIOSH shiftwork booklet
- Sleep Enhancement Training System (Experimental)
  Interventions: Behavioral: Sleep Enhancement Training System

INTERVENTIONS:
Behavioral: Sleep Enhancement Training System — 4 week program of readings and relaxation programs
  Arms: Sleep Enhancement Training System
Behavioral: NIOSH shiftwork booklet — weekly readings about coping with shiftwork
  Arms: NIOSH shiftwork booklet

SUMMARY:
The purpose of this study is to determine if a modified version of the Sleep Enhancement Fatigue Reduction Training (SEFRT) system can improve sleep and health-related symptoms and quality of life in shiftwork-naive new nurse graduates.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking nurses scheduled to work at least 2 consecutive night shifts per week in the next 2 months

Exclusion Criteria:

* > 6 months experience working night-shift
* current diagnosis of sleep disorder or affective illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
actigraphy measures of sleep | 6 weeks

SECONDARY OUTCOMES:
subjective measures of sleep and well-being | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R Alsten, PhD, Principal Investigator — Inner Health, Inc.
Locations (1):
- University of California, San Francisco, San Francisco, California, United States